CLINICAL TRIAL: NCT00272285
Title: A Double-blind, Randomized, Parallel, Comparative Study to Evaluate the Efficacy and Safety of Ramosetron Plus Dexamethasone Injection for the Prevention of Chemotherapy-Induced Vomiting and Nausea
Brief Title: A Study of Ramosetron Plus DX, Dexamethasone, Compared to Granisetron Plus DX for the Prevention of Vomiting and Nausea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06003/TnIO01
Record Dates: First submitted 2006-01-03; First posted 2006-01-05 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Vomiting; Nausea
Keywords: Serotonin antagonists; Randomized controlled trial; Combination drug therapy; Double-blind method
MeSH Terms: conditions — Vomiting; Nausea | interventions — ramosetron; Granisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intravenous (IV)
  Interventions: Drug: Ramosetron
- 2 (Active Comparator): Intravenous (IV)
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Ramosetron — IV, concomitant administration with dexamethasone
  Arms: 1
Drug: Granisetron — IV, concomitant administration with dexamethasone
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ramosetron plus dexamethasone injection with granisetron plus dexamethasone injection for the prevention of chemotherapy-induced vomiting and nausea.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age between 20-74 years old (inclusive) of either sex
* Cancer subject is scheduled to receive the designated chemotherapy programs
* Subject without symptoms of vomiting for at least one week before dosing trial medication
* Subject with ECOG performance status scale no greater than 2
* Subject has signed the written informed consent form

Exclusion Criteria:

* Subject has received radiotherapy to the abdomen or pelvis within 4 weeks before entering this study
* Subject has received the designated chemotherapy programs within 6 months before entering the study
* Subject has known heart failure or myocardial infraction or with laboratory abnormalities at screening
* Subject has known concurrent diseases that may cause vomiting
* Subject has taken medications that could influence the outcome of the study within 3 days before entering the study
* Subject with a history of allergy or intolerance to ramosetron, granisetron or dexamethasone
* Female subject who is pregnant or breastfeeding
* Subject with life expectancy less than 3 months
* Subject participated other investigational drug trial within 1 month before entering this study

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without vomiting after the start of chemotherapy for 24 hours | 1 Day

SECONDARY OUTCOMES:
Response rate of vomiting prevention | 1 Day
The number of vomiting episodes | 1 Day
The nausea degree evaluated by patient's 10-cm visual analogue scale (VAS) | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Use central contact, Study Chair — Astellas Pharma Inc
Locations (2):
- Taiwan (2):
  - Tainan
  - Taipei

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=150